CLINICAL TRIAL: NCT00159510
Title: A Controlled Prospective Randomized Open-Label Study of Methylene Blue and Inhaled Nitric Oxide in Patients With Septic Shock and Acute Lung Injury
Brief Title: Studies of Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome
Acronym: MB-NO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit the patients due to the short supply and changed local hospital protocol
Sponsor: Northern State Medical University (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Prof., Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4001.721.132; Helse Nord (Norway), project (Other: HelseNord); number 4001.721.132 (Other: HelseNord)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Sepsis
Keywords: sepsis, methylene blue, nitric oxide, acute lung injury
MeSH Terms: conditions — Sepsis; Acute Lung Injury | interventions — Methylene Blue; Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): The control group with neither nitric oxide nor methylene blue used
- MB alone (Active Comparator): Single methylene blue used
  Interventions: Drug: Methylene blue
- NO alone (Active Comparator): Nitric oxide alone used
  Interventions: Drug: Nitric oxide
- MB+NO (Active Comparator): Both nitric oxide and methylene blue used
  Interventions: Drug: Methylene blue & nitric oxide

INTERVENTIONS:
Drug: Methylene blue — Injection bolus of 2 mg/kg PBW and infusion of 0.2 mg/kg/hr
  Arms: MB alone
Drug: Nitric oxide — An inhalation of NO via ETT at 10 ppm, partially weaned by 72 hrs of therapy
  Other Names: Not actual
  Arms: NO alone
Drug: Methylene blue & nitric oxide — See the dosage in the previous arms
  Other Names: Not actual
  Arms: MB+NO

SUMMARY:
Nitric oxide (NO) plays a pivotal role in maintenance of normal vascular tone. However, in sepsis the excessive production of NO results in myocardial depression, vasoplegia, and cytotoxic effects, thus promoting shock and multiple organ dysfunction. A recently completed study from our group showed advantageous cardiovascular effects of continuously infused methylene blue (MB), an inhibitor of NO pathway, in human septic shock. In another investigation, we have found that the combination of inhaled NO and continuously infused MB attenuates endotoxin-induced acute lung injury (ALI) in sheep. Our intention is, in a new study, to test the hypothesis that the combination of MB and NO (MB+NO) improves both cardiovascular and pulmonary functions as well as clinical outcome in patients with septic shock and ALI. Forty mechanically ventilated patients diagnosed with hyperdynamic septic shock and ALI, will be randomized to groups receiving

1. Conventional treatment (control group)(n =10);
2. MB infusion in addition to conventional treatment (n=10);
3. Inhaled NO in addition to conventional treatment (n=10);
4. MB infusion combined with inhaled NO (MB+NO) in addition to conventional treatment (n=10).

DETAILED DESCRIPTION:
The therapy with either MB+NO or NO or MB alone will be prolonged for up to 24 h or until resolution of septic shock, whichever occurs first. MB will be injected as a bolus of 2 mg/kg subsequently followed by dose-titrated infusion. The latter beginning with 0.25 mg/kg/h continuing within the range of from 0.05 to 0.5 mg/kg/h. The goal is to maintain mean arterial pressure within the range of 70-90 mm Hg, with the purpose of reducing any concurrent vasopressor therapy. The NO therapy will be started from 10 ppm and aimed at maintaining the mean pulmonary artery pressure at the lowest possible levels by inhaling NO in concentrations from 1 to 20 ppm.

ELIGIBILITY:
Inclusion Criteria:

1. Informed written consent from the patient, or a written consent from a relative together with a the doctor responsible for the treatment of the patient
2. Aged 18 years or above.
3. Severe sepsis diagnosed less than 72 h prior to randomization.
4. Septic shock defined as a syndrome characterized by severe sepsis in association with either:

   * a MAP <70 mm Hg for at least 30 consecutive minutes despite fluid resuscitation or,
   * a requirement for vasopressor support with a constant dose rate of either epinephrine >0,05 mcg/kg/min and/or norepinephrine >0.05 mcg/kg/min and/or dopamine >5 mcg/kg/min and/or phenylephrine >0.5 mcg/kg/min for at least 30 consecutive minutes to maintain a MAP >90 mm Hg
5. Cardiac index (CI) must be >3.5 l/min/m2, pulmonary artery occlusion pressure (PAOP) must be between 8 and 18 mm Hg, and in the opinion of the investigator the patient must be adequately fluid resuscitated
6. A 4 French Pulsiocath thermodilution catheter (Pulsion Medical Systems, München, Germany) in place in one of the femoral arteries and a 7 French thermistor-tipped balloon floatation catheter (Swan Ganz) in the pulmonary artery for determination of hemodynamics, including extravascular lung water index (EVLWI).
7. A dedicated intravenous line for infusion of MB
8. A respirator with a device for delivery of gaseous NO to the inspiration gas and equipped with analysis tools for lung mechanics
9. The patients will be treated in intensive care units with the possibility to provide full life support for the whole duration of the study
10. In female patients a negative pregnancy test will be requires before inclusion unless the patient is either in the post-partum period or known to have undergone prior tubal ligation or hysterectomy, or be postmenopausal

Exclusion Criteria:

* 1) Patients who have received vasopressor infusion therapy as described in the definition of septic shock either intermittently or continuously for a period of more than 24 h prior to randomization 2) The use of any vasoactive drug infusion other than epinephrine, norepinephrine, dopamine, phenylephrine and dobutamine, at the time of study entry 3) Patients in whom either vasodilators or dobutamine are contraindicated 4) Patients who cannot have their MAP managed safely within the range of 70-90 mm Hg (e.g. patients with raised intracranial pressure) 5) Shock due to any cause other than severe sepsis (e.g. drug reaction or drug overdose, adrenal insufficiency, pulmonary embolus, burn injury etc.) 6) Patients that are immunocompromised due to any of the following:
* known corticosteroid therapy either greater than or equal to a total daily dose equivalent to 1 mg/kg or greater than 70 mg/day of oral prednisolone for at least 7 consecutive days within one month prior to study entry,
* clinically suspected or known to have Acquired Immunodeficiency Syndrome (AIDS),
* granulocyte count less than 1000/mm3 due to a cause other than severe sepsis (e.g. metastatic or hematological malignancies or chemotherapy),
* immunosuppressant therapy (e.g. due to an organ or bone marrow transplant), 7) Underlying disease, exclusive of septic shock, which is expected to cause death within 1 month from study entry 8) Within 30 days prior to this study, the patient should not have been included in any other randomized therapeutic study of an agent not licensed, or administration of any other investigational agent for the treatment of sepsis and/or septic shock. Patients must not participate in such studies for at least 30 days after enrolment into this study.

  9) Pregnant women, pregnancy test required of any fertile women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 28
  Mortality rate by Day 28

SECONDARY OUTCOMES:
Duration of inotropic and vasopressor support | 7 Days
  Duration of vasopressor and/or inotrope suppor
Severity of organ dysfunction | 7 Days
  Number of organ-specific dysfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, MD, PhD, Principal Investigator — Northern State Medical University
Locations (1):
- University Hospital #1, Arkhangelsk, Russia, Russia